CLINICAL TRIAL: NCT05193747
Title: The Depth of Paediatric Anaesthesia: Observational Trial
Acronym: ANAPED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, Clinical Professor, Brno University Hospital
Other Study IDs: KDAR ANADEPTH 2022
Record Dates: First submitted 2022-01-02; First posted 2022-01-18 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Anesthesia Awareness
Keywords: Anesthesia; Awareness; Pediatric; Children
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paediatric patients scheduled for general anesthesia: Paediatric patients (between 1 year -19 years) undergoing elective general anaesthesia with presumed duration over 1 hour will be eligible for inclusion
  Interventions: Other: Anesthesia depth monitoring

INTERVENTIONS:
Other: Anesthesia depth monitoring — BIS monitor will be placed on the forehead according to the manufacturer recommendation and the anaesthesia team will be blinded to BIS monitor during the whole case. The initial BIS tracing will be recorded starting the surgery initiation (defined as the depth of anesthesia by the anaesthesiologist to initiate surgical intervention) and ending with end of surgical intervention.

SUMMARY:
Perioperative measurement of the Depth of anaesthesia is currently recommended part of daily anaesthesia good clinical practice. The optimal depth of anaesthesia measured by Bispectral index could be between 40-60. The lower (over 60) depth of anaesthesia could be associated with accidental intraoperative episodes of awareness and deeper (below 40) anaesthesia could lead to higher adverse events or even haemodynamic instability.

DETAILED DESCRIPTION:
The hypothesis of the trial is that during the perioperative period serious fluctuations outside the recommended target depth of anaesthesia could occur. These fluctuations and the cumulative time spent in the shallow (over 60 BIS) or deep (under 40 BIS) could be associated with postoperative complications like emergence delirium (PAED over 10, and PAED over 12- 2 measurement methods), postoperative nausea and vomiting (PONV) and other postoperative complications (respiratory, hemodynamic).

Paediatric patients (between 1 year -19 years) undergoing elective general anaesthesia with presumed duration over 1 hour will be eligible for inclusion. The patients will be screened for eligibility during the preanaesthesia visit in the anaesthesiology examination room. After the Ethics committee and registration of the study at clinicaltrials.gov, the patients will be enrolled - according to the trial design. There is a presumption that informed consent won't be needed for participation due to observational trial. The anaesthesia induction will be performed either inhalation or intravenous route. After anaesthesia induction BIS monitor will be placed on the forehead according to the manufacturer recommendation and the anaesthesia team will be blinded to BIS monitor during the whole case. The initial BIS tracing will be recorded starting the surgery initiation (defined as the depth of anesthesia by the anaesthesiologist to initiate surgical intervention) and ending with end of surgical intervention. The incidence of periods outside the recommended anaesthesia depth will be recorded (episode is defined by ≥ 30 seconds interval outside the predefined limits, the end of episode is defined by the return to recommended BIS level). The cumulative time spent outside the recommended BIS levels will be evaluated as the primary outcome measure. The anaesthesiologist's ability to respond to fluctuations defined as YES / NO response, type of intervention and latency of the anaesthesiologist's response to fluctuation will be evaluated. The BIS recording will be terminated at the time the surgical intervention is finished. After surgery/anaesthesia, the patient will be transferred to ICU or post-anaesthesia care unit (PACU), where the incidence of emergence delirium (defined by PEAD score over 10 and over 12 - according to 2 measurement methods) and the incidence of PONV will be recorded. Also, cumulative incidence of overall complication in the postoperative period (desaturation, the need for oxygen therapy, haemodynamic instability, arrhythmias (over 150/min, below 50/min, allergic reactions) will be recorded. In the case of a critical BIS value (≥90, ≤10), blinding will be interrupted due to patient safety and the value will be notified to the anesthesiology team and the event will be recorded as a critical event.

ELIGIBILITY:
Inclusion Criteria:

* Age 1 year-19 years
* Elective general anaesthesia with presumed duration over 60 minutes
* BIS monitor available

Exclusion Criteria:

* Outside the age limits
* Acute surgery
* Presumed anaesthesia duration below 1 hour
* Without the possibility of BIS monitoring
* Patient indicated for sedation and mechanical ventilation after anesthesia

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Paediatric patients (between 1 year -19 years) undergoing elective general anaesthesia with presumed duration over 1 hour will be eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Cumulative time outside recommended BIS levels | intraoperatively
  The cumulative time spent outside the recommended BIS levels will be evaluated
Periods outside recommended BIS levels | intraoperatively
  The incidence of periods outside the recommended anaesthesia depth will be recorded (episode is defined by ≥ 30 seconds interval outside the predefined limits, the end of episode is defined by the return to recommended BIS level).

SECONDARY OUTCOMES:
Ability to respond | Intraoperatively
  The anaesthesiologist's ability to respond to fluctuations defined as YES / NO response, type of intervention and latency of the anaesthesiologist's response to fluctuation will be evaluated.
Incidence of emergence delirium | 2 hours postoperatively
  After surgery/anaesthesia, the patient will be transferred to ICU or PACU, where the incidence of emergence delirium (defined by PEAD over 10 and over 12 - 2 measurement methods) and the incidence of PONV will be recorded.
Incidence of overall complications | 2 hours postoperatively
  Cumulative incidence of overall complication in the postoperative period (desaturation, the need for oxygen therapy, haemodynamic instability, arrhythmias (over 150/min, below 50/min, allergic reactions) will be recorded.
Delay to respond | Intraoperatively
  Latency of the anaesthesiologist's response to fluctuation - defined in seconds from the onset of fluctuation to the end of fluctuation = return to the recommended BIS level
Incidence of postoperative nausea and vomiting (PONV( | 2 hours postoperatively
  Incidence of PONV at PACU

CONTACTS AND LOCATIONS:
Overall Officials: Petr Stourac, prof. MD., Ph.D., MBA, Study Chair — Department of paediatric anaesthesia and intensive care medicine
Locations (1):
- Brno University Hospital, Brno, South Moravian, Czechia

IPD SHARING:
Plan to Share IPD: Undecided